CLINICAL TRIAL: NCT04104360
Title: Impact of Galacto-oligosaccharides on the Intestinal Microbial Composition and -Activity: a Proof of Concept Study
Brief Title: Galacto-oligosaccharides and Intestinal Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 18-039
Record Dates: First submitted 2019-09-17; First posted 2019-09-26 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Healthy Adults
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Galacto-oligosacchardies (Experimental): During this period subjects will receive 7.2 grams of Vivinal GOS supplements three times daily for four weeks
  Interventions: Dietary Supplement: Galacto-oligosaccharides
- Maltodextrin (Placebo Comparator): During this period subjects will receive 7.2 grams of maltodextrin three times daily for four weeks
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Galacto-oligosaccharides — During this period subjects will receive 7.2 grams of Vivinal GOS supplements three times daily for four weeks
  Arms: Galacto-oligosacchardies
Dietary Supplement: Maltodextrin — During this period subjects will receive 7.2 grams of maltodextrin supplements three times daily for four weeks
  Arms: Maltodextrin

SUMMARY:
Dietary intake of galacto-oligosaccharides (GOS) may have beneficial effects on host health by affecting the microbiota composition and -activity. So far studies focused on analyses in fecal samples, while the primary site of carbohydrate fermentation is the proximal colon. To date, no studies have been performed in humans on the more proximal microbiota and the impact of fermentable carbohydrates. Further insights on the more proximal colonic microbiota would aid to targeted approaches to improve intestinal health. Therefore, we aim to study the effect of GOS on the intestinal microbiota composition and -activity in healthy adults, by sampling the more proximal human colon in a physiological condition. The primary objective of this study is to investigate the impact of four weeks GOS supplementation on intestinal microbiota composition and -activity, by sampling the proximal part of the human colon in a physiological condition. Furthermore, this study has four secondary objectives: First, to compare the intestinal microbiota composition and -activity of the proximal colon vs. distal colon at baseline and after four weeks GOS supplementation. Second, compare the luminal microbiota composition vs. mucosa adherent microbiota composition of the proximal vs. distal colon at baseline and after four weeks GOS supplementation. Third, monitor the effects of four weeks GOS supplementation on gastrointestinal symptoms. The study conforms to a randomized, double-blind, placebo-controlled, parallel design. Study population includes healthy human volunteers (male and female), 18-50 years of age. One intervention arm will include 7.2 grams of Vivinal® GOS Powder three times daily for four weeks. The other intervention arm subjects will receive placebo product (7.2 grams maltodextrin) three times daily for four weeks. At the start and end of the intervention period, several measurements will take place. The main study parameter is the change in microbial composition and -activity induced by GOS intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Based on medical history no gastrointestinal complaints can be defined.
2. Regular stool frequency ranging from 3 times/day - 3 times/week.
3. Body Mass Index (BMI) ≥ 20 and < 30 kg/m2.
4. Weight-stable for at least 90 days prior to participation (no change in bodyweight, i.e. < 3kg).
5. Willing to be informed in case of unexpected findings.

Exclusion Criteria:

1. History of any disease or surgery interfering with the study aims, limiting participating or completing the study protocol.
2. Self-admitted human immunodeficiency virus-positive state.
3. Disease with a life expectancy shorter than 5 years.
4. Abdominal surgery interfering with gastrointestinal function, upon judgment of the medical doctor, who will decide on in- or exclusion based on the surgery applied.
5. Use of antibiotics within 90 days prior to the study.
6. Use of anticoagulation medication (except Ascal).
7. Use of proton pump inhibitors.
8. Use of other medication will be reviewed by a medical doctor, who will decide on in- or exclusion based on the drug(s) used.
9. Last colonoscopy within 90 days prior to the study.
10. Inadequate or painful (self-reported) colonoscopy undergone in the past.
11. American Society of Anesthesiologists (ASA) classification > 2.
12. Smoking.
13. Pregnancy or lactation.
14. Plan to lose weight or follow a specific diet within the study period.
15. Alcohol intake >14 units/week.
16. Use of laxatives within 14 days prior to the study.
17. Drug use.
18. Administration of probiotic or prebiotic supplements, investigational drugs or participation in any scientific intervention study, which may interfere with this study (to be decided by the principle investigator), in the 14 days prior to the study.
19. History of side effects towards intake of prebiotic supplements.
20. Self-admitted lactose intolerance.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Microbial composition, as determined by state of the art (e.g. HiSeq) sequencing of 16S rRNA genes in colonic luminal/fecal samples and biopsies. | Change from baseline to four weeks supplementation
  Total DNA will be extracted from fecal, small intestinal fluid and biopsy samples using the repeated bead-beating method. This method has been optimized and standardized for the extraction of total bacterial DNA from human fecal samples. Isolated DNA will be used for amplification of the V4 region of the collective 16S rRNA genes using barcoded primers, while fecal and intestinal DNA as target. Afterwards, the NG-Tax pipeline will be used for microbiota profiling. A variety of programs, such as R, and in house scripts will be used for bioinformatics analyses and multivariate statistics.
Microbial activity as determined by metatranscriptomics using RNA in colonic luminal samples and biopsies. | Change from baseline to four weeks supplementation
  Microbiota activity profiling will be performed by metatranscriptomics. In short, RNA will be isolated from the luminal samples, followed by removal of rRNA and subsequent conversion of residual RNA into cDNA. The cDNA will serve as target for paired-end HiSeq sequencing. Obtained sequence reads will be phylogenetically and functionally annotated as described before. Dedicated R-scripts as well as programs such as iPath will be used for bioinformatic analyses, including metabolic mapping, and interpretation to determine which bacterial group is performing what activities. In addition, key metabolites of saccharolytic and protein fermentation (such as (branched) chain fatty acids) will be assessed by High-performance liquid chromatography (HPLC).

CONTACTS AND LOCATIONS:
Overall Officials: D. Keszthelyi, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No